CLINICAL TRIAL: NCT05099107
Title: COMPIS- Congenital Myopathy Intervention Study. An Open-label, Cross Over, Randomised, Controlled Study Using Oral Salbutamol
Brief Title: Changes of Motor Function Tests in Congenital Myopathy Subjects Treated With Oral Salbutamol as Compared to no Treatment
Acronym: COMPIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: COMPIS; 2019-001147-51 (EudraCT Number)
Record Dates: First submitted 2021-10-15; First posted 2021-10-29 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-03

CONDITIONS: Congenital Myopathy; Neuromuscular Diseases; Musculoskeletal Diseases; Nemaline Myopathy; Centronuclear Myopathy; Myosin Storage Myopathy
Keywords: oral salbutamol; motor function measure 32
MeSH Terms: conditions — Myotonia Congenita; Neuromuscular Diseases; Musculoskeletal Diseases; Myopathies, Nemaline; Myopathies, Structural, Congenital; Muscular Dystrophy, Emery-Dreifuss | interventions — Albuterol; Tablets; Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): congenital myopathy patients in this group will receive daily oral salbutamol, three times daily.
  Interventions: Drug: Salbutamol (as Salbutamol Sulfate) 2 Mg Oral Tablet; Drug: Salbutamol Only Product in Oral Dose Form
- Non treatment (No Intervention): Congenital myopathy patients in this group will not receive any salbutamol nor placebo.

INTERVENTIONS:
Drug: Salbutamol (as Salbutamol Sulfate) 2 Mg Oral Tablet — taken 3 times daily for 6 months
  Other Names: Ventolin tablet
  Arms: Treatment
Drug: Salbutamol Only Product in Oral Dose Form — taken 3 times daily for 6 months
  Other Names: Ventolin oral syrup
  Arms: Treatment

SUMMARY:
Congenital myopathies (CM) is a large group of muscle disorders, presenting with hypotonia and non-progressive generalised muscle weakness, which can lead to motor developmental delay.More than 20 genes can cause CM and currently there is no curative treatment for this disorder.

Case reports and a smaller study have previous reported that oral salbutamol has benefited subjects with different types of congenital myopathies by increasing their muscle strength.The exact effect of salbutamol in muscle cells isn't exactly known but it has been hypothesized to have an anabolic effect by triggering different pathways inside the muscle cells which increase cell proliferation, decrease apoptosis, decreases proteolysis and increases protein synthesis.

The aim of our study is evaluate if daily oral salbutamol can increase the muscle function and muscle strength in these patients after 6 months on treatment, compared to no treatment.

DETAILED DESCRIPTION:
We hypothesise that congenital myopathy subjects treated with daily oral salbutamol will increase in their motor function measure 32 test (MFM32) with at least 3 points after 6 months of treatment as compared to no treatment. We have calculated that a sample size of 18 subjects is needed for this study.

Congenital myopathy subjects will be recruited from the whole of Sweden and the study will be performed at the Sahlgrenska university hospital in Gothenburg Sweden.

The subjects must have clinical symptoms consistent with congenital myopathy and have a verified mutation in a gene known to cause congenital myopathy.

After a screening period of 6 months the eligible subjects will be randomised into two groups, group A and group B . During period 1, group A will receive oral salbutamol 3 times daily and the group B will have no treatment.They will be evaluated after 6 months. Then after a washout period of 1 month, Period 2 will begin where the groups will cross-over, i.e group A will have no treatment and group B will receive oral salbutamol 3 times daily.

In total each subject will be evaluated 5 times during 19 months with the same battery of muscle function and strength tests performed each time.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from legal guardians/patients and patient (where applicable)
* Subject must have a confirmed congenital myopathy(CM) diagnosis defined as:

  * Clinical symptoms consistent with CM with pathohistological findings on muscle biopsy and known genetic mutation consistent with CM OR
  * Clinical symptoms consistent with CM with unspecific pathohistological changes but known genetic mutation consistent with CM
* Stabile motor function tests over at least 6 months (between baseline and screening)
* If on other medications- stabile dose for at least 6 months prior to start
* At least 1 point on Motor function measure 32 test is (MFM32) at screening visit.

>5- <31 years of age (from 6 years to 30 years of age)

* Women of fertile age must be on oral contraceptives
* Underwent cardiac evaluation with ECG and 2D echocardiography in the last 2 years and has no signs or symptoms of cardiac abnormality.

Exclusion Criteria:

* Subject with clinical symptoms consistent with CM but has no confirmed genetic mutation and only unspecific changes on muscle biopsy that are not confined to just CM but can be seen in other disorders.
* Younger than 6 years of age and older than 30 years
* Subject receives 94 or more points on MFM32 test at screening visit.
* Subject doesn't not speak Swedish and a translator is needed in order to perform the tests included in the study.
* Subject smokes more than 10 cigarettes a day or has smoked more than 10 cigarettes in the last year
* Subject has tracheostomy
* Subject receives no points on motor function measure test at screening
* Subject has other concomitant chronic diagnosis that can affect the patients motor function, in the opinion of the investigator
* Subject is currently or has been on oral corticosteroids in the last 6 months
* Subject has arrhythmia as seen on electrocardiogram(ECG), confirmed by cardiologist
* Subject has cardiomyopathy as seen on ultrasound, confirmed by cardiologist
* Subject has severe behavioural and/ cognitive problems that preclude participation in the study, in the opinion of the investigator
* Subject is allergic or hypersensitive to study drug or any of its constituents
* Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow- up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator;
* Subject is currently taking any other investigational drug or has taken any other investigational drug within 3 months prior to the first dose of study medication
* Subject is planning on participating in any other study during the duration of this study.
* Female subjects of fertile age that are or are planning to become pregnant during the study.
* Female subjects that have given birth up to 1 year prior to baseline visit and/or are nursing up to 1 month prior of baseline visit
* Subject has a fracture in the last 6 months before the study start or has acquired a fracture during the study.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Motor function measure test 32 (MFM32) | 19 months
  score presented as a total score from 0 to 96 points, the higher the score the better motor function

SECONDARY OUTCOMES:
timed function tests | 5 evaluations in 19 months
  seconds
6 minute walk test | 5 evaluations in 19 months
  meters/minute for speed calculation, as well as total distance walked.
hand grip test | 5 evaluations in 19 months
  measured in pounds
5 consecutive 9 hole PEG test | 5 evaluations in 19 months
  measured in seconds
muscle myometry test using a hand held myometer | 5 evaluations in 19 months
  measured in newtons
Activity limitation ACTIVLIM- quality of life questionnaire | 5 evaluations in 19 months
  measured as total score, 0-32 max points, the higher the score the less the limitation in activities

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Darin, M.D, Principal Investigator — Vastra Gotaland Region
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data(IPD) that underlie results in a publication
Time Frame: The data will be available starting 6 months after publication